CLINICAL TRIAL: NCT02067455
Title: This is a Non-randomized, Single-center, Prospective Investigation on Exercise Capacities of Left Ventricular Assist Devices Recipients
Brief Title: REVADE : Right Ventricular Function and Exercise in Left Ventricular Assist Device Patients : Echocardiographic Study
Acronym: REVADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-A01798-37; 35RC13_8808_REVADE (Other: Rennes University Hospital)
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Left Ventricular Assist Devices Patients
Keywords: Right ventricular function; echocardiography; left ventricular assist device; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LVAD patients (Other)
  Interventions: Other: adding 2 cardiopulmonary exercise testings : peak oxygen consumption (VO2 max) and stress echocardiography

INTERVENTIONS:
Other: adding 2 cardiopulmonary exercise testings : peak oxygen consumption (VO2 max) and stress echocardiography
  Other Names: - resting echocardiography; - routine bloods tests; - 1 stress echocardiography on a supine bicycle over the follow; - 1 peak oxygen consumption recorded while breathing through a gas analyser

SUMMARY:
Heart failure is a public health problem, responsible for 150.000 admissions, 32.000 deaths, 1% of public health expenditure each year in France. Heart transplantation remains the standard of care in patients for which medical therapy is not sufficient. But heart transplantation is a limited resource, as a result of donor shortages. It is therefore possible to consider mechanical circulatory support for patients awaiting heart transplantation or for those who are not suitable for transplantation. Left Ventricular Assist Devices (LVAD) are portable pumps which help the left side of the heart to provide appropriate "cardiac" output. in this type of device, right heart is not assisted and must work on its own, LVADs are thus implanted in patients whose right ventricular function is normal.

The aim of the REVADE study is to assess right ventricular echocardiographic parameters in this population, especially on physical exercise, for a better understanding of right ventricular adaptation to this long-term modified pressure pattern.

DETAILED DESCRIPTION:
This is a non-randomized, single-center, prospective investigation on exercise capacities of LVAD recipients.

LVAD patients already have in our unit the following regular monitoring:

* clinical examination
* Minnesota Living with Heart Failure Questionnaire (MLHFQ)
* SF-36 Health Survey
* Six-Minute Walk Test
* resting echocardiography
* routine blood tests.

The REVADE pilot study consists in adding 2 cardiopulmonary exercise testings to their existing follow-up : peak oxygen consumption (VO2 max) and stress echocardiography.

We plan to do 1 stress echocardiography on a supine bicycle over the follow-up, and 1 peak oxygen consumption recorded while breathing through a gas analyzer.

Total study length of time will be 1 year. Expected number of enrolled patients is 18.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular assist device (LVAD) recipients
* age > 18 years
* able to give consent

Exclusion Criteria:

* adults legally protected (under judicial protection, guardianship, or supervision) or deprived of liberty
* patients unable to provide sufficient effort for exercise testing
* poor echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
assessment of right chambers dimensions for the evaluation of right ventricular function | 12 months
assessment of RV strain for the evaluation of right ventricular function | 12 months
assessment of RV shortening fraction for the evaluation of right ventricular function | 12 months
assessment of TAPSE for the Evaluation of right ventricular function | 12 months
assessment of RV fractional Area change for the evaluation of right ventricular function | 12 months
assessment of Tricuspid annulus tissue doppler imaging for the evaluation of right ventricular function | 12 months
Tricuspid regurgitation analysis for the evaluation of right ventricular function | 12 months
pulmonary pressures analysis for the evaluation of right ventricular function | 12 months
Assessment of RV strain rate for the evaluation of right ventricular function | 12 months

SECONDARY OUTCOMES:
peak oxygen consumption (VO2 max) as a functional evaluation of VO2 max on exercise | 12 months
quality of life scores as an assessment of quality of life | 12 months
BNP levels as an assessment of BNP levels | 12 months
Blood pressure monitoring as an assessment of blood pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Erwan DONAL, Principal Investigator — Rennes University Hospital; ERWAN FLECHER, Principal Investigator — Rennes University Hospital
Locations (1):
- Service de cardiologie - Rennes university hospital, Rennes, France

REFERENCES:
- [Derived] Aymami M, Donal E, Guihaire J, Le Helloco A, Federspiel M, Galli E, Carre F, Lelong B, Chabanne C, Corbineau H, Leguerrier A, Verhoye JP, Flecher E. Rest and Exercise Adaptation of the Right Ventricular Function in Long-Term Left Ventricular Assist Device Patients: A Prospective, Pilot Study. J Card Fail. 2016 Mar;22(3):240-1. doi: 10.1016/j.cardfail.2015.12.009. Epub 2015 Dec 17. No abstract available. PMID 26705752